CLINICAL TRIAL: NCT00403481
Title: A Prospective, Open Label, Single Arm Study to Evaluate the Safety and Efficacy of an Olmesartan Medoxomil Based Treatment Regimen in Type II Diabetic Patients With Hypertension
Brief Title: An Examination of the Blood Pressure Lowering Ability and Safety of Olmesartan Medoxomil in Patients With Type II Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: William Waverczak, Daiichi Sankyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 866-449
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Results first posted 2009-09-15 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin Receptor Blocker; Calcium Channel Blocker; Angiotensin Converting Enzyme Inhibitor; Hydrochlorothiazide; Stage I and II Hypertension; Type II Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

ARMS (1):
- Active treatment (Experimental): Blood pressure (BP) measurements were taken every three weeks for 12 weeks. In accordance with their BP results, participants either stayed on their current medication or were started on the next higher regimen at the 3, 6, or 9 week visits. All participants began at 20 mg olmesartan, once daily for 3 weeks. The next higher regimen was olmesartan 40 mg, followed by olmesartan 40 mg + 12.5 mg hydrochlorothiazide, followed by olmesartan 40 mg + 25 mg of hydrochlorothiazide.
  Interventions: Drug: olmesartan medoxomil; Drug: Olmesartan medoxomil plus Hydrochlorothiazide

INTERVENTIONS:
Drug: olmesartan medoxomil — Olmesartan medoxomil tablets, once daily
Drug: Olmesartan medoxomil plus Hydrochlorothiazide — Olmesartan medoxomil and hydrochlorothiazide combination tablets, once daily, if necessary

SUMMARY:
This study will examine the ability of olmesartan medoxomil to lower the blood pressure of patients with Type II diabetes and high blood pressure. The medication being tested has been approved by the FDA for the treatment of high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type II diabetes that are on stable treatment with hypoglycemic agents
* Patients with a mean seated systolic blood pressure (MSSBP) greater than or equal to 140 mmHg but <200 mmHg and a MSDBP less than or equal to 114 mmHg following a 3 to 4-week single-blind placebo run-in period
* The difference in MSSBP between Visits 3 and 4 or between Visits 4 and 4X must be less than or equal to 10 mmHg
* Patients with a mean daytime (8AM - 4PM) SBP > 130 mmHg and less than or equal to 199 mmHg and a mean daytime DBP less than or equal to 114 as measured by an ambulatory blood pressure monitoring device (ABPM) following placebo run-in period
* If female, must have negative serum pregnancy test at screening and be either post-menopausal, had a hysterectomy or tubal ligation at least 6 months before consent or if of childbearing potential, must practice approved measures of birth control throughout study

Exclusion Criteria:

* History of stroke or transient ischemic attack (TIA) within the last one year
* History of myocardial infarction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, and/or unstable angina pectoris within the past 6 months
* Presence of overt proteinuria at screening
* Severe hypertension (DBP greater than or equal to 115 mmHg or SBP greater than or equal to 200 mmHg)
* Patients with secondary hypertension of any etiology, such as renal disease, pheochromocytoma, or Cushing's syndrome
* Type I or Type II diabetes requiring insulin
* Evidence of symptomatic resting bradycardia, congestive heart failure, or hemodynamically significant cardiac valvular disease
* Presence of heart block greater than first degree sinoatrial block, Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial fibrillation, or Atrial Flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Searcy, Arkansas
  - Los Angeles, California
  - Roseville, California
  - Tustin, California
  - DeLand, Florida
  - Pembroke Pines, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - Madisonville, Kentucky
  - Auburn, Maine
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Jackson, Mississippi
  - Florissant, Missouri
  - Williamsville, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - New Talenwell, Tennessee
  - New Tazewell, Tennessee
  - Colleyville, Texas
  - Corpus Christi, Texas
  - Richardson, Texas
  - Murray, Utah
  - Norfolk, Virginia

REFERENCES:
- [Derived] Kereiakes DJ, Neutel JM. Seated cuff blood pressure-lowering efficacy of an olmesartan medoxomil-based treatment regimen in patients with type 2 diabetes mellitus. Drugs R D. 2011 Sep 1;11(3):251-7. doi: 10.2165/11592830-000000000-00000. PMID 21777013
- [Derived] Neutel JM, Kereiakes DJ; BENIFICIARY Investigators. An olmesartan medoxomil-based treatment algorithm is effective in achieving 24-hour BP control in patients with type 2 diabetes mellitus, regardless of age, race, sex, or severity of hypertension: subgroup analysis of the BENIFICIARY study. Am J Cardiovasc Drugs. 2010;10(5):289-303. doi: 10.2165/11584690-000000000-00000. PMID 20712386
- [Derived] Neutel JM, Kereiakes DJ, Waverczak WF, Stoakes KA, Xu J, Shojaee A. Effects of an olmesartan medoxomil based treatment algorithm on 24-hour blood pressure control in patients with hypertension and type 2 diabetes. Curr Med Res Opin. 2010 Mar;26(3):721-8. doi: 10.1185/03007990903553556. PMID 20085534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 24 US sites over 10 months from November 2006 to August 2007 from each physician's clientele base. Approximately 200 eligible subjects, men and women at least 18 years of age with stage I/II hypertension and stable type 2 diabetes mellitus, were to be enrolled on active treatment.
Pre-assignment Details: 192 participants started this single arm titration study. Participants remained in their group or were titrated at 3-week intervals depending on achievement their blood pressure goals.
Groups:
- Active Treatment Period: All participants started this arm with 20 mg olmesartan medoxomil (Olm). After 3 weeks participants were titrated to 40g Olm, if their blood pressure was not controlled. After 6 weeks they were titrated to the next step which now included Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg if their blood pressure was not controlled. After 9 weeks they were titrated to the next step which now included Olm + HCTZ 25 mg if their blood pressure was not controlled.
Period: Olmesartan Medoxomil (Olm) 20 mg
Arm/Group | Active Treatment Period
Started | 192
Completed | 186
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1
Period: Olm 40 mg
Arm/Group | Active Treatment Period
Started | 182 (186 -4 met their blood pressure goal (remained on olmesartan 20 mg) = 182)
Completed | 177
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Period: Olm 40 mg + Hydrochlorothiazide 12.5 mg
Arm/Group | Active Treatment Period
Started | 173 (177 -4 met their blood pressure goal (remained on olmesartan 40 mg)= 173)
Completed | 168
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Period: Olm 40 mg + Hydrochlorothiazide 25 mg
Arm/Group | Active Treatment Period
Started | 144 (168 -24 met their blood pressure goal (remained on olmesartan 40 mg/hydrochlorothiazide 12.5mg)= 144)
Completed | 142
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Treatmant Arm: All participants started this arm with 20 mg olmesartan medoxomil (Olm). After 3 weeks participants were titrated to 40g Olm, if their blood pressure was not controlled. After 6 weeks they were titrated to the next step which now included Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg if their blood pressure was not controlled. After 9 weeks they were titrated to the next step which now included Olm + HCTZ 25 mg if their blood pressure was not controlled.
Arm/Group | Active Treatmant Arm
Number analyzed (Participants) | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 107
Race/Ethnicity, Customized [Number; unit: Participants]
  Black/African American | 43
  Asian | 3
  White | 145
  Native Hawaiian/Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 192
Diastolic BP [Mean (Standard Deviation); unit: mm Hg] | 90.0 (10.0)
Heart rate [Mean (Standard Deviation); unit: beats/min] | 76.4 (10.4)
Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 158.1 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Systolic BP (SBP) as Measured by 24-hour ABPM.
Description: Participants had a 24-hour ambulatory blood pressure session at baseline and after 12 weeks of treatment. This outcome measure pooled all participants regardless of their titration history during the study.
Time Frame: baseline and 12 weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 172
mm Hg | -20.4 (0.88)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, One-sample t-test — No multiplicity adjustments

2. Secondary Outcome: Change From Baseline to Week 12 in Mean Daytime and Nighttime Ambulatory Blood Pressure Measurement (Systolic).
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 172
mm Hg
  Daytime | -22.3 (1.05)
  Nighttime | -18.8 (0.94)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, one-sample t-test — <0.0001 for both daytime and nighttime. No multiplicity adjustments

3. Secondary Outcome: Change From Baseline to Week 12 in Ambulatory BP Measurement (Systolic)During the Last 2 Hours of the Last (Week 12) 24-hour Dosing Period.
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM. Of the 172 ABPM participants, only 169 had the required measurements for this outcome analysis.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 169
mm Hg | -18.6 (1.11)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, One-sample t-test

4. Secondary Outcome: Change From Baseline to Week 12 in Ambulatory BP Measurement (Systolic)During the Last 4 Hours of the Last (Week 12 ) 24-hour Dosing Period.
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM.Of the 172 ABPM participants, only 171 had the required measurements for this outcome analysis.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 171
mm Hg | -18.2 (1.00)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p = 0.0001, one-sample t-test — No multiplicity adjustments

5. Secondary Outcome: Change From Baseline to Week 12 in Ambulatory BP Measurement (Systolic)During the Last 6 Hours of the Last (Week 12 ) 24-hour Dosing Period.
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM. Of the 172 ABPM participants, only 171 had the required measurements
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 171
mm Hg | -18.6 (0.92)

6. Secondary Outcome: Change From Baseline to Week 12 in Mean 24-hour Ambulatory BP (Diastolic)
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 172
mm Hg | -11.1 (0.54)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, one-sample t-test

7. Secondary Outcome: Change in Daytime and Nighttime Ambulatory Blood Pressure (Diastolic) From Baseline to Week 12
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 172
mm Hg
  Daytime | -12.0 (0.68)
  Nighttime | -10.2 (0.55)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, one-sample t-test — <0.0001 applies to both the daytime and nighttime analyses

8. Secondary Outcome: Change in Ambulatory Blood Pressure (Diastolic) From Baseline to Week 12 During the Last 2 Hours of the Last (Week 12 ) 24-hour Dosing Period.
Description: as for outcome 1
Time Frame: baseline and 12 Weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM.Of the 172 participants, only 169 had the required measurements for this outcome analysis.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 169
mm Hg | -10.6 (0.78)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, one-sample t-test

9. Secondary Outcome: Change in Ambulatory BP (Diastolic) From Baseline to Week 12 During the Last (Week 12 ) 4 and 6 Hours of the Last 24-hour Dosing Period.
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: A total of 192 participants started. Eighteen dropped out. All Ambulatory Blood Pressure Monitoring (ABPM) Subjects (N=172) consisted of all subjects in the efficacy cohort who had a baseline and week 12 ABPM. Of the 172 ABPM participants, only 171 had the required measurements for this outcome analysis.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Overall Study Population
Number analyzed (Participants) | 171
mm Hg
  4 hours | -10.7 (0.66)
  6 hours | -10.8 (0.61)
Statistical Analysis 1: Comparison: Overall Study Population; Test type: Superiority or Other; p < 0.0001, one-sample t-test — <0.0001 applies to both 4 hour and 6 hour analyses

ADVERSE EVENTS:
Time Frame: 12 week treatment period plus 30 days after the last dose of study medication.
Description: Safety assessments included physical examination, reporting of adverse events, and changes in laboratory values. At each visit, the investigator determined whether any adverse events had occurred by evaluating the subject. Subjects were to be questioned in a general way, without asking about the occurrence of any specific symptoms.
Groups:
- Olmesartan 20 mg; Olmesartan 40 mg; Olmesartan 40 mg and Hydrochlorothiazide 12.5 mg; Olmesartan 40 mg and Hydrochlorothiazide 25 mg: All participants started with 20 mg olmesartan medoxomil (Olm). After 3 weeks participants were titrated to 40g Olm, if their blood pressure was not controlled. After 6 weeks they were titrated to the next step which now included Olm 40 mg + hydrochlorothiazide (HCTZ) 12.5 mg if their blood pressure was not controlled. After 9 weeks they were titrated to the next step which now included Olm + HCTZ 25 mg if their blood pressure was not controlled.
Arm/Group | Olmesartan 20 mg | Olmesartan 40 mg | Olmesartan 40 mg and Hydrochlorothiazide 12.5 mg | Olmesartan 40 mg and Hydrochlorothiazide 25 mg
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/182 | 1/173 | 0/144
Other Adverse Events (participants affected / at risk) | 4/192 | 5/182 | 3/173 | 6/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan 20 mg (N=192) | Olmesartan 40 mg (N=182) | Olmesartan 40 mg and Hydrochlorothiazide 12.5 mg (N=173) | Olmesartan 40 mg and Hydrochlorothiazide 25 mg (N=144)
Death due to arteriosclerotic cardiovascular disease (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan 20 mg (N=192) | Olmesartan 40 mg (N=182) | Olmesartan 40 mg and Hydrochlorothiazide 12.5 mg (N=173) | Olmesartan 40 mg and Hydrochlorothiazide 25 mg (N=144)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 3
Bronchitis (Infections and infestations) | 3 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If identified by Daiichi Sankyo Inc., any of DSI's confidential information, as defined to the author, shall be deleted. Nothing in our site agreement shall be taken as giving Daiichi Sankyo, Inc. any right of editorial control over any publication prepared by the study site.